CLINICAL TRIAL: NCT04568525
Title: Microwave Radiation for Early Diagnostics of Pneumonia in Patients With COVID-19
Brief Title: Passive Microwave Radiometry (MWR) and AI for COVID-19 Complications Early Diagnostics of Lungs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyrgyz State Medical Academy (Other)
Collaborators: University of Edinburgh (Other); IMU University, Malaysia (Other)
Responsible Party: Principal Investigator, Batyr Osmonov, Head of respiratory department, Kyrgyz State Medical Academy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 01-2/141 27
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: CT - scan; X-Ray; MWR
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized clinical trials
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COVID - 19 patients (Active Comparator)
  Interventions: Diagnostic Test: Passive Microwave Radiometry
- COVID - 19 and pneumonia patients (Active Comparator)
  Interventions: Diagnostic Test: Passive Microwave Radiometry
- Health patients (Active Comparator)
  Interventions: Diagnostic Test: Passive Microwave Radiometry

INTERVENTIONS:
Diagnostic Test: Passive Microwave Radiometry — The MWR2020 (ormer RTM-01-RES) device is a unique commercially available CE marked device. It is registered in UK MHRA MDN 40802 as Microwave thermography system for clinical studies. The device is already registered in Kyrgyzstan for breast cancer diagnostics. During the 1980-90s there were several works on identification of excess of microwave emission due to fluid in lungs (on phantoms) which could be indication of inflammatory, process, cancer and other lung disorders.Later results were confirmed by clinical studies for lung cancer

SUMMARY:
World Health Organization (WHO) declared COVID-19 it as a global pandemic. It becomes clear that the virus spreading mostly deadly due to limited to access to diagnostics tests and equipment. Traditional radiography and CT remain the main methods of the initial examination of the chest organs. Now, most of the diagnostics has been focused on PCR, chest x-Ray/CT manifestations of COVID-19. However, there are problems with CT due to infection control issues, the inefficiencies introduced in CT room decontamination, and lack of CT availability in LMIC (Low Middle Income Countries). Passive microwave radiometry (MWR) is a cheap, non-radioactive and portable technology. It has already been used for diagnostics of cancer, and other diseases. The investigators have tested if MWR could be used for early diagnostics of pulmonary COVID-19 complications.

This was a randomized controlled trial (195 subjects) to evaluate the effectiveness of diagnostics using MWR in patients with pneumonia caused by COVID-19 while they are in hospitals of Kyrgyzstan, and healthy individuals.

The investigator have measured skin (IR) and internal (MWR) temperature by recording passive electromagnetic radiation through the chest wall in the projection of the lungs at 30 symmetrical points on both sides. Pneumonia and lung damage were diagnosed by X-RAY/CT scan and doctor's final diagnosis (pn+/pn-). COVID-19 was determined by PCR test (covid+/covid-).

Overall, the study suggests that the use of MWR is a convenient and safe method for screening diagnostics in COVID-19 patients with suspected pneumonia. Since MWR is an inexpensive, it will ease the financial burden for both patients and the countries, especially in LMIC

ELIGIBILITY:
Inclusion Criteria:

* Male and female gender, age 18-75 years
* Positive RT-PCR result of COVID-19
* Place of birth and residence (<800m above sea level)
* Informed consent

Exclusion Criteria:

* - Lack of fever in a healthy group
* Exacerbation of COPD, very severe COPD with hypoxia (FEV1 <40%, saturation <92% at an altitude of 760 m).
* Co-morbidities, such as cardiovascular diseases, i.e. unstable systemic arterial hypertension, coronary heart disease; stroke; sleep apnea; pneumothorax last 2 months.
* Neurological, rheumatological or psychiatric illnesses, including excessive smoking (> 20 cigarettes per day)
* Kidney failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 50/50
Enrollment: 195 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Determine sensitivity and specificity of MWR diagnostics of pneumonia in patients with COVID-19. (diagnosed by PCR and CT) | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Educational - clinical - scientific medical center of KSMA, Bishkek, Chui, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sahu KK, Mishra AK, Lal A. Comprehensive update on current outbreak of novel coronavirus infection (2019-nCoV). Ann Transl Med. 2020 Mar;8(6):393. doi: 10.21037/atm.2020.02.92. PMID 32355837
- [Background] Lu R, Zhao X, Li J, Niu P, Yang B, Wu H, Wang W, Song H, Huang B, Zhu N, Bi Y, Ma X, Zhan F, Wang L, Hu T, Zhou H, Hu Z, Zhou W, Zhao L, Chen J, Meng Y, Wang J, Lin Y, Yuan J, Xie Z, Ma J, Liu WJ, Wang D, Xu W, Holmes EC, Gao GF, Wu G, Chen W, Shi W, Tan W. Genomic characterisation and epidemiology of 2019 novel coronavirus: implications for virus origins and receptor binding. Lancet. 2020 Feb 22;395(10224):565-574. doi: 10.1016/S0140-6736(20)30251-8. Epub 2020 Jan 30. PMID 32007145
- [Background] Wu D, Wu T, Liu Q, Yang Z. The SARS-CoV-2 outbreak: What we know. Int J Infect Dis. 2020 May;94:44-48. doi: 10.1016/j.ijid.2020.03.004. Epub 2020 Mar 12. PMID 32171952
- [Background] Liu K, Chen Y, Lin R, Han K. Clinical features of COVID-19 in elderly patients: A comparison with young and middle-aged patients. J Infect. 2020 Jun;80(6):e14-e18. doi: 10.1016/j.jinf.2020.03.005. Epub 2020 Mar 27. PMID 32171866
- [Background] Zhong Z, Hu Y, Yu Q, Li Y, Li P, Huang W, Liu J, Liu J, Xie X, Zhao W. Multistage CT features of coronavirus disease 2019. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2020 Mar 28;45(3):250-256. doi: 10.11817/j.issn.1672-7347.2020.200144. Chinese, English. PMID 32386015
- [Derived] Osmonov B, Ovchinnikov L, Galazis C, Emilov B, Karaibragimov M, Seitov M, Vesnin S, Losev A, Levshinskii V, Popov I, Mustafin C, Kasymbekov T, Goryanin I. Passive Microwave Radiometry for the Diagnosis of Coronavirus Disease 2019 Lung Complications in Kyrgyzstan. Diagnostics (Basel). 2021 Feb 7;11(2):259. doi: 10.3390/diagnostics11020259. PMID 33562419